CLINICAL TRIAL: NCT01005888
Title: LEVP2005-1/Part B: A Double-blind, Placebo-Controlled, Clinical Study to Investigate the Efficacy and Safety of Purified C1 Esterase Inhibitor (Human) as Prophylactic Treatment to Prevent HAE Attacks
Brief Title: C1 Esterase Inhibitor (C1INH-nf) for the Prevention of Acute Hereditary Angioedema (HAE) Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LEVP2005-1/Part B
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Results first posted 2010-06-03 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; HAE; C1 esterase inhibitor (human); C1INH-nf
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C1INH-nf First, then Placebo (Experimental): 1,000 Units (U) of C1INH-nf administered intravenously (IV) every 3 to 4 days (approximately twice weekly) for 12 weeks, followed by matching placebo (saline) administered IV every 3 to 4 days for 12 weeks.
  Interventions: Biological: C1 esterase inhibitor [human] (C1INH-nf); Drug: Placebo (saline)
- Placebo First, then C1INH-nf (Experimental): Matching placebo (saline) administered IV every 3 to 4 days (approximately twice weekly) for 12 weeks, followed by 1,000 U of C1INH-nf administered IV every 3 to 4 days for 12 weeks.
  Interventions: Biological: C1 esterase inhibitor [human] (C1INH-nf); Drug: Placebo (saline)

INTERVENTIONS:
Biological: C1 esterase inhibitor [human] (C1INH-nf)
Drug: Placebo (saline)

SUMMARY:
The study objective was to determine the safety and efficacy of C1INH-nf for the prevention of acute HAE attacks.

DETAILED DESCRIPTION:
Subjects were given diary cards and instructed to document all HAE attacks on a daily basis. Subjects evaluated their symptoms over the previous 24 hours, noting the severity and duration of swelling at each of 5 locations (abdominal, genitourinary, facial, respiratory [including laryngeal], and/or extremity).

The study design also allowed for administration of open-label C1INH-nf (1,000 U of C1INH-nf administered IV [repeated after 60 minutes, if necessary] for treatment of laryngeal angioedema or if deemed necessary by the investigator; 1,000 U of C1INH-nf administered IV [single dose] prior to emergency surgical procedures).

A total of 26 subjects were enrolled in the study. One subject received open-label C1INH-nf but withdrew prior to randomization. Another subject was randomized but withdrew prior to receiving study drug. Twenty-four (24) subjects were randomized and treated with blinded study drug. In total, 25 subjects received at least 1 dose of study drug and were analyzed for safety; all 25 subjects were exposed to C1INH-nf and 23 subjects were exposed to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Documented HAE
* Normal C1q level
* Relatively frequent angioedema attacks (at least 2 per month on average)

Exclusion Criteria:

* Low C1q level
* B-cell malignancy
* Presence of anti-C1INH autoantibody
* History of allergic reaction to C1INH or other blood products
* Narcotic addiction
* Current participation in any other investigational drug study or within the past 30 days
* Participation in a C1 esterase inhibitor trial, or received blood or a blood product in the past 90 days
* Pregnancy or lactation
* Any clinically significant medical condition, such as renal failure, that in the opinion of the investigator would interfere with the subject's ability to participate in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-03-14 (Actual); Primary Completion 2007-08-22 (Actual); Study Completion 2007-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (16):
- United States (16):
  - Allergy and Immunology Associates, Scottsdale, Arizona
  - University of California, San Diego, San Diego, California
  - Allergy and Asthma Clinical Research, Inc, Walnut Creek, California
  - Atlanta Allergy and Asthma Clinic, Suwanee, Georgia
  - Hawaii Pacific Health Research Institute, Honolulu, Hawaii
  - Welborn Clinic Allergy and Immunology, Evansville, Indiana
  - Lake Charles Memorial Hospital, Lake Charles, Louisiana
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Libby Clinic, Libby, Montana
  - Mount Sinai School of Medicine, New York, New York
  - Nationwide Childrens Hospital Clinical Research, Columbus, Ohio
  - Allergy Clinic of Tulsa, Tulsa, Oklahoma
  - Allergy Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - AARA Research Center, Dallas, Texas
  - Tyler County Hospital, Woodville, Texas
  - St. Joseph's Hospital/Cornerstone Healthcare, Parkersburg, West Virginia

REFERENCES:
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Lumry WR, Miller DP, Newcomer S, Fitts D, Dayno J. Quality of life in patients with hereditary angioedema receiving therapy for routine prevention of attacks. Allergy Asthma Proc. 2014 Sep-Oct;35(5):371-6. doi: 10.2500/aap.2014.35.3783. PMID 25295804
- [Derived] Lumry W, Manning ME, Hurewitz DS, Davis-Lorton M, Fitts D, Kalfus IN, Uknis ME. Nanofiltered C1-esterase inhibitor for the acute management and prevention of hereditary angioedema attacks due to C1-inhibitor deficiency in children. J Pediatr. 2013 May;162(5):1017-22.e1-2. doi: 10.1016/j.jpeds.2012.11.030. Epub 2013 Jan 11. PMID 23312695
- [Derived] Zuraw BL, Busse PJ, White M, Jacobs J, Lumry W, Baker J, Craig T, Grant JA, Hurewitz D, Bielory L, Cartwright WE, Koleilat M, Ryan W, Schaefer O, Manning M, Patel P, Bernstein JA, Friedman RA, Wilkinson R, Tanner D, Kohler G, Gunther G, Levy R, McClellan J, Redhead J, Guss D, Heyman E, Blumenstein BA, Kalfus I, Frank MM. Nanofiltered C1 inhibitor concentrate for treatment of hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):513-22. doi: 10.1056/NEJMoa0805538. PMID 20818886

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 26 subjects were enrolled in the study (see Detailed Description). One subject received open-label C1 esterase inhibitor (C1INH-nf) but withdrew prior to randomization. Another subject was randomized but withdrew prior to receiving study drug. 24 subjects were randomized and began therapy with blinded study drug in Period 1.
Period: First Intervention
Arm/Group | C1INH-nf First, Then Placebo | Placebo First, Then C1INH-nf
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Period: Second Intervention
Arm/Group | C1INH-nf First, Then Placebo | Placebo First, Then C1INH-nf
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- C1INH-nf First, Then Placebo: 1,000 U of C1INH-nf administered IV every 3 to 4 days (approximately twice weekly) for 12 weeks, followed by matching placebo (saline) administered IV every 3 to 4 days for 12 weeks.
- Open-label C1INH-nf Only: One subject received open-label C1INH-nf but withdrew prior to randomization.
- Randomized, Not Treated: One subject was randomized but withdrew prior to receiving study drug.
- Total: Total of all reporting groups
Arm/Group | C1INH-nf First, Then Placebo | Placebo First, Then C1INH-nf | Open-label C1INH-nf Only | Randomized, Not Treated | Total
Number analyzed (Participants) | 12 | 12 | 1 | 1 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 0 | 1 | 5
  Between 18 and 65 years | 9 | 10 | 1 | 0 | 20
  >=65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 1 | 0 | 22
  Male | 3 | 0 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Hereditary Angioedema (HAE) Attacks During Each Prophylactic Therapy Period
Description: An HAE attack was defined as the subject-reported indication of swelling at any location following a report of no swelling on the previous day. Analyses include observed attack counts and normalized attack counts (i.e., the number of attacks observed during each therapy period, normalized for the number of days the subject participated in that period).
Time Frame: 12 weeks
Population: The Efficacy Dataset (N=22) consisted of all randomized subjects who completed 12 weeks of therapy in Period 1 and received at least one infusion of study drug in Period 2.
Measure: Mean (Standard Deviation); unit: attacks
Groups:
- C1INH-nf: 1,000 U of C1INH-nf administered IV every 3 to 4 days (approximately twice weekly) for 12 weeks.
- Placebo: Matching placebo (saline) administered IV every 3 to 4 days (approximately twice weekly) for 12 weeks.
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 22 | 22
attacks
  Observed | 6.1 (5.43) | 12.7 (4.80)
  Normalized | 6.3 (5.54) | 12.7 (4.65)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA — Observed number of attacks
Statistical Analysis 2: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA — Normalized number of attacks

2. Secondary Outcome: Number of Subject Withdrawals During Each Prophylactic Therapy Period
Description: At the end of each therapy period, each subject was assigned a yes/no drop-out status. A drop-out was defined as a subject who did not have a Week 12 visit record.
Time Frame: 12 weeks
Population: The Safety Dataset (N=24) consisted of all randomized subjects who received at least 1 complete or partial infusion of study drug. 24 subjects began Period 1 (12 C1INH-nf, 12 placebo) and received study drug. 22 subjects crossed over to Period 2 (11 placebo, 11 C1INH-nf) and received study drug. Thus, 23 randomized subjects received each therapy.
Measure: Number; unit: participants
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 23 | 23
participants
  Period 1 | 1 | 1
  Period 2 | 1 | 1
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p > 0.999, Fisher Exact — Period 1
Statistical Analysis 2: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p > 0.999, Fisher Exact — Period 2

3. Secondary Outcome: Average Severity of HAE Attacks During Each Prophylactic Therapy Period
Description: All attacks in each therapy period were assigned a value of 1 (mild), 2 (moderate), or 3 (severe). Attack severity was considered the highest value assigned by the subject to any swelling location during the attack. Average severity was set to 0 if there was no attack in a period.
Time Frame: 12 weeks
Population: Efficacy Dataset.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale | 1.3 (0.85) | 1.9 (0.35)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0008, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Average Duration of HAE Attacks During Each Prophylactic Therapy Period
Description: The duration of an attack was measured from the first report of swelling at any one of the five locations (abdominal, genitourinary, facial, respiratory [including laryngeal], or extremity) until the first subsequent report of "no swelling" at all five locations.
Time Frame: 12 weeks
Population: Efficacy Dataset.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 22 | 22
days | 2.1 (1.13) | 3.4 (1.39)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Open-label C1INH-nf Infusions Required During Each Prophylactic Therapy Period
Description: The study design allowed for subjects to be treated with open-label C1INH-nf for laryngeal angioedema, if deemed necessary by the investigator, or prior to emergency surgical procedures.
Time Frame: 12 weeks
Population: Efficacy Dataset.
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 22 | 22
infusions | 4.7 (8.66) | 15.4 (8.41)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: Total Number of Days of Swelling During Each Prophylactic Therapy Period
Description: A day of swelling was defined as a day that a subject reported swelling at any of the five locations (abdominal, genitourinary, facial, respiratory [including laryngeal], or extremity).
Time Frame: 12 weeks
Population: Efficacy Dataset.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 22 | 22
days | 10.1 (10.73) | 29.6 (16.90)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Antigenic C1 Inhibitor (C1INH) Serum Levels
Description: Change in antigenic C1INH serum levels from pre-infusion to 1 hour post-infusion at Visit 1 and Weeks 4, 8, and 12. Pre-infusion samples obtained at Visit 1 of each therapy period (i.e., baseline) were used to determine change at 1 hour post-infusion for all visits.
Time Frame: Pre-infusion to 1 hour post-infusion at Visit 1 and Weeks 4, 8, and 12
Population: Efficacy Dataset subjects with data at both sampling time points (N=19 C1INH-nf, N=22 placebo).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 19 | 22
mg/dL
  Visit 1 pre-infusion | 14.3 (15.08) | 14.2 (14.71)
  Visit 1 change at 1 hour post-infusion | 7.9 (3.70) | -0.1 (2.17)
  Week 4 change at 1 hour post-infusion | 9.8 (5.08) | 0.1 (5.04)
  Week 8 change at 1 hour post-infusion | 7.2 (5.62) | -0.3 (3.08)
  Week 12 change at 1 hour post-infusion | 8.4 (5.93) | 1.1 (5.98)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Visit 1 change at 1 hour post-infusion
Statistical Analysis 2: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Week 4 change at 1 hour post-infusion
Statistical Analysis 3: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney) — Week 8 change at 1 hour post-infusion
Statistical Analysis 4: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0028, Wilcoxon (Mann-Whitney) — Week 12 change at 1 hour post-infusion

8. Secondary Outcome: Functional C1INH Serum Levels
Description: Percent change in functional C1INH serum levels from pre-infusion to 1 hour post-infusion at Visit 1 and Weeks 4, 8, and 12. Pre-infusion samples obtained at Visit 1 of each therapy period (i.e., baseline) were used to determine change at 1 hour post-infusion for all visits. Functional C1INH serum levels are expressed as a percent of total detectable C1INH (i.e., functional C1INH/total detectable C1INH).
Time Frame: Pre-infusion to 1 hour post-infusion at Visit 1 and Weeks 4, 8, and 12
Population: Efficacy Dataset subjects with data at both sampling time points (N=20 C1INH-nf, N=22 placebo).
Measure: Mean (Standard Deviation); unit: percent of functional C1INH
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 20 | 22
percent of functional C1INH
  Visit 1 pre-infusion | 33.9 (17.21) | 31.7 (21.54)
  Visit 1 percent change at 1 hour post-infusion | 32.0 (18.95) | -2.4 (9.41)
  Week 4 percent change at 1 hour post-infusion | 36.6 (17.62) | 5.3 (26.16)
  Week 8 percent change at 1 hour post-infusion | 32.1 (19.08) | 5.4 (15.74)
  Week 12 percent change at 1 hour post-infusion | 33.9 (21.07) | 0.8 (23.92)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Visit 1 percent change at 1 hour post-infusion
Statistical Analysis 2: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Week 4 percent change at 1 hour post-infusion
Statistical Analysis 3: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Week 8 percent change at 1 hour post-infusion
Statistical Analysis 4: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney) — Week 12 percent change at 1 hour post-infusion

ADVERSE EVENTS:
Time Frame: Up to 6 months (i.e., 24 weeks) of therapy and 3 months of follow-up. 25 subjects received at least 1 dose of study drug and were analyzed for safety; all 25 were exposed to C1INH-nf and 23 were exposed to placebo (see Detailed Description).
Description: Presented are treatment-emergent adverse reactions considered to be related to study drug. There were no serious adverse reactions considered related to study drug.
Arm/Group | C1INH-nf | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 3/25 | 0/23
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C1INH-nf (N=25) | Placebo (N=23)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to sponsor for pre-review. If sponsor requests, PI must delete sponsor confidential information before publication and/or delay publication for 90 days so sponsor can file for patents or take other action to protect its patent rights.